CLINICAL TRIAL: NCT03255707
Title: A Comparative Study Between Dissociative Treatment and Binocular Interactive Treatment in Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Suha Ahmed Amin, Ophthalmology Specialist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 293/2016
Record Dates: First submitted 2017-08-06; First posted 2017-08-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Amblyopia
Keywords: Amblyopia; Interactive Binocular Treatment; Dissociative Treatment; Occlusion; Patching
MeSH Terms: conditions — Amblyopia; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Patients of the study will be recruited from the ophthalmology outpatient clinic of Ain Shams University Hospital.100 patients of both sexes with amblyopia will be enrolled. Informed consents will be obtained from adult patients and children's parents.
  Patients will be assigned randomly:
  Group A:50 patients will receive the gold standard occlusion therapy while playing a video game (Lazy Eye Tetris games such as Lazy Eye Blocks ®).Group B:50 patients will receive dichoptic treatment in the form of playing a video game (Lazy Eye Tetris games such as Lazy Eye Blocks ®) while wearing a red/green goggle.Each group will be subdivided according to age:
  1)4 to 7 years. 2)>7 to 12 years. 3)>12 to 30 years.
  Hours of occlusion /dichoptic treatment will be classified according to the degree of amblyopia:
  * Mild to moderate amblyopia (Best corrected visual acuity (BCVA)< 0.2) : 2-4 hours
  * Severe (BCVA> 0.2) : 4-6 hours
  All patients will undergo full ophthalmological examination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): 50 patients will receive the gold standard occlusion therapy
  Interventions: Device: eye patch
- Group B (Experimental): 50 patients will receive dichoptic treatment in the form of playing a video game (Lazy Eye Blocks ®) while wearing a red/green goggle.
  Interventions: Device: dichoptic treatment

INTERVENTIONS:
Device: eye patch — Occluding the better seeing eye for a given number of hours daily
  Arms: Group A
Device: dichoptic treatment — dichoptic treatment in the form of playing a video game (Lazy Eye Blocks ®) while wearing a red/green goggle.
  Arms: Group B

SUMMARY:
Amblyopia is a unilateral or, infrequently, a bilateral reduction of best corrected visual acuity which cannot be attributed to coexisting eye or visual pathway disease. Amblyopia can be due to eye-crossing occurring in early childhood or due to error of refraction whether a high difference between the two eyes or very high bilateral refractive errors.Another cause could be visual deprivation like the presence of congenital cataract.

The prevalence of amblyopia worldwide is approximately 1%-5% .In Egypt, a study that was held in Upper Egypt, found that the prevalence of amblyopia was 1.49%, which is higher in rural areas than in urban areas.

Several modalities of treatment for amblyopia are available, yet occlusion treatment is the gold standard involving covering the good eye with a patch for a prescribed period of time ranging from 10 minutes daily to all waking hours. However, its effectiveness decreases in older children and adults.

Disadvantages include prolonged treatment leading to poor compliance, patching related distress, relationship strain and stigma. In extreme cases, non-compliance with patching results in a costly hospital admission to supervise the patching treatment. In addition, wearing a patch eliminates any advantage of binocularity. Not to mention that not all patients respond to patching and of those who do, many have residual amblyopia after treatment is stopped regardless of compliance. More importantly, binocular vision is not automatically restored once the vision in the amblyopic eye has been improved. In fact, once the patch is removed after therapy, the amblyopic eye could be suppressed by the better seeing eye and can lose some of the gains achieved as a result of therapy.

Another modality of treatment is atropine eye drops and optical penalisation which are usually secondary treatments to failed patching but carrying the same disadvantages as the ordinary patching.

Advances in amblyopia treatment include dichoptic training, perceptual learning, and video gaming. These depend on the fact that the adult brain has been shown to be much more plastic than it was once believed to be and hence have the advantage of expanding the age of response in adults.

Perceptual learning approaches have the advantage of being a dichoptic (binocular treatment using both eyes) approach which is independent of age and type of amblyopia.

A step further to conventional treatment is the use of a home-based approach allowing remote internet monitoring of treatment between office visits and hence better compliance. In addition a video game version of the treatment is developed to make it more enjoyable for improving compliance.

Our goal is to compare the outcome between the gold standard occlusion therapy and one of the dichoptic treatments.

DETAILED DESCRIPTION:
Introduction Amblyopia is a unilateral or, infrequently, a bilateral reduction of best corrected visual acuity which cannot be attributed to coexisting eye or visual pathway disease. Amblyopic eyes may have decreased contrast sensitivity and accommodation deficit. The fellow eye is not often normal but has subtle deficits.This can be explained by interocular suppression, or inhibition of the amblyopic eye by the strong eye, with psychophysical and physiological evidence.

Amblyopia can be classified as follows: 1) Strabismic occurring in early childhood 2) Refractive: a) Anisometropic b) High bilateral refractive errors 3) Visual deprivation.

The prevalence of amblyopia worldwide is approximately 1%-5%. In Egypt, a study that was held in Upper Egypt, found that the prevalence of amblyopia was 1.49%, which is higher in rural areas than in urban areas.

Several modalities of treatment for amblyopia are available, yet occlusion treatment is the gold standard involving covering the good eye with a patch for a prescribed period of time ranging from 10 minutes daily to all waking hours. However, its effectiveness decreases in older children and adults.

Disadvantages include prolonged treatment leading to poor compliance, patching related distress, relationship strain and stigma. In extreme cases, non-compliance with patching results in a costly hospital admission to supervise the patching treatment. In addition, wearing a patch eliminates any advantage of binocularity. Not to mention that not all patients respond to patching and of those who do, many have residual amblyopia after treatment is stopped regardless of compliance. More importantly, binocular vision is not automatically restored once the vision in the amblyopic eye has been improved. In fact, once the patch is removed after therapy, the amblyopic eye could be suppressed by the better seeing eye and can lose some of the gains achieved as a result of therapy.

Another modality of treatment is atropine eye drops and optical penalisation which are usually secondary treatments to failed patching but carrying the same disadvantages as the ordinary patching.

Advances in amblyopia treatment include dichoptic training, perceptual learning, and video gaming. These depend on the fact that the adult brain has been shown to be much more plastic than it was once believed to be and hence have the advantage of expanding the age of response in adults.

Perceptual learning approaches have the advantage of being a dichoptic (binocular treatment) approach which is independent of age and type of amblyopia. Furthermore, it has been shown recently that therapy promotes binocular vision by strengthening stereopsis and reducing suppression.

A step further to conventional treatment is the use of a home-based approach allowing remote internet monitoring of treatment between office visits and hence better compliance. In addition a video game version of the treatment is developed to make it more enjoyable for improving compliance.

Aim of the work:

To compare the gold standard occlusion therapy alone with dichoptic therapy

Patients and Methods:

Design:

The study will be a prospective experimental controlled study.

Patients of the study:

From the vicinity of the ophthalmology outpatient clinic of Ain Shams University Hospital, 100 patients of both sexes with amblyopia will be enrolled to this study. Informed consents will be obtained from adult patients and children's parents.

Patients will be assigned randomly into two groups:

Group A: 50 patients will receive the gold standard occlusion therapy

Group B: 50 patients will receive dichoptic treatment in the form of playing a video game (Lazy Eye Blocks ®) while wearing a red/green goggle.

Each group will be subdivided according to age:

1. From 4 to 7 years.
2. From above 7 to 12 years.
3. From above 12 to 30 years.

Hours of occlusion will be classified according to the degree of amblyopia:

* Mild to moderate amblyopia (Best corrected visual acuity (BCVA)< 0.2): 2-4 hours occlusion
* Severe (BCVA> 0.2): 4-6 hours occlusion

Hours of dichoptic treatment in group B will be classified according to the degree of amblyopia:

* Mild to moderate amblyopia (BCVA< 0.2): 2-4 hours of treatment
* Severe (BCVA> 0.2): 4-6 hours of treatment

Methods

All patients will undergo the following:

1. Full medical and ophthalmic history
2. Examination:

A) External Appearance:

Anomalous Head Position, globes (e.g., proptosis), lids (e.g. ptosis).

B) Refraction:

With and without cyclopegia

C) Visual acuity:

With and without correction using Snellen acuity chart and preferential looking test for non-verbal patients.

D) Motility:

Ductions and versions (9 positions of gaze) E) Angle of deviation if any

F) Fixation :

Fixation behavior (fixation preference) will be tested via base down 10 prism diopter fixation preference test.

G) Quantitative Binocular vision assessment H) Anterior segment examination. I) Posterior segment examination using indirect ophthalmoscopy with a 20 diopter lens through a dilated pupil.

All patients in Group A will receive the gold standard occlusion therapy. All patients in Group B will receive dichoptic treatment

ELIGIBILITY:
Inclusion Criteria:

* Any degree of amblyopia
* Orthotropia in primary position.

Exclusion Criteria:

* Any ocular disease affecting vision
* Angle of deviation in primary position (Heterotropia)
* Adult patients and children's parents unwilling to enter or complete the study
* Ignorance of patients to use the video game

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
visual acuity | 6 months
  Best corrected visual acuity in the amblyopic eye

SECONDARY OUTCOMES:
Compliance | 6 months
  Compliance of the patient to treatment
crowding ratio | 6 months
  crowded vs uncrowded visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Hazem H Nouh, MD, Study Chair — Ophthalmology department, faculty of medicine, Ain Shams University; Mohammad A Rashad, MD, Study Chair — Ophthalmology department, faculty of medicine, Ain Shams University; Walid M El-Zawahry, MD, Study Director — Ophthalmology department, faculty of medicine, Ain Shams University; Ahmad T Ismail, MD, Study Director — Ophthalmology department, faculty of medicine, Ain Shams University; Suha A Hussein, M.Sc, Principal Investigator — Ophthalmology department, faculty of medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals (Demerdash), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldebasi YH. Prevalence of amblyopia in primary school children in Qassim province, Kingdom of Saudi Arabia. Middle East Afr J Ophthalmol. 2015 Jan-Mar;22(1):86-91. doi: 10.4103/0974-9233.148355. PMID 25624680
- [Background] Attebo K, Mitchell P, Cumming R, Smith W, Jolly N, Sparkes R. Prevalence and causes of amblyopia in an adult population. Ophthalmology. 1998 Jan;105(1):154-9. doi: 10.1016/s0161-6420(98)91862-0. PMID 9442792
- [Background] Birch EE. Amblyopia and binocular vision. Prog Retin Eye Res. 2013 Mar;33:67-84. doi: 10.1016/j.preteyeres.2012.11.001. Epub 2012 Nov 29. PMID 23201436
- [Background] Ding J, Klein SA, Levi DM. Binocular combination in abnormal binocular vision. J Vis. 2013 Feb 8;13(2):14. doi: 10.1167/13.2.14. PMID 23397039
- [Background] Ding J, Levi DM. Rebalancing binocular vision in amblyopia. Ophthalmic Physiol Opt. 2014 Mar;34(2):199-213. doi: 10.1111/opo.12115. Epub 2014 Jan 12. PMID 24417338
- [Background] Dixon-Woods M, Awan M, Gottlob I. Why is compliance with occlusion therapy for amblyopia so hard? A qualitative study. Arch Dis Child. 2006 Jun;91(6):491-4. doi: 10.1136/adc.2005.090373. Epub 2006 Mar 10. PMID 16531452
- [Background] Fu J, Li SM, Liu LR, Li JL, Li SY, Zhu BD, Li H, Yang Z, Li L, Wang NL; Anyang Childhood Eye Study Group. Prevalence of amblyopia and strabismus in a population of 7th-grade junior high school students in Central China: the Anyang Childhood Eye Study (ACES). Ophthalmic Epidemiol. 2014 Jun;21(3):197-203. doi: 10.3109/09286586.2014.904371. Epub 2014 Apr 17. PMID 24742059
- [Background] Ganekal S, Jhanji V, Liang Y, Dorairaj S. Prevalence and etiology of amblyopia in Southern India: results from screening of school children aged 5-15 years. Ophthalmic Epidemiol. 2013 Aug;20(4):228-31. doi: 10.3109/09286586.2013.809772. PMID 23865603
- [Background] He HY, Hodos W, Quinlan EM. Visual deprivation reactivates rapid ocular dominance plasticity in adult visual cortex. J Neurosci. 2006 Mar 15;26(11):2951-5. doi: 10.1523/JNEUROSCI.5554-05.2006. PMID 16540572
- [Background] Hess RF, Babu RJ, Clavagnier S, Black J, Bobier W, Thompson B. The iPod binocular home-based treatment for amblyopia in adults: efficacy and compliance. Clin Exp Optom. 2014 Sep;97(5):389-98. doi: 10.1111/cxo.12192. Epub 2014 Aug 18. PMID 25131694
- [Background] Hess RF, Mansouri B, Thompson B. Restoration of binocular vision in amblyopia. Strabismus. 2011 Sep;19(3):110-8. doi: 10.3109/09273972.2011.600418. PMID 21870914
- [Background] Levi DM, Li RW. Perceptual learning as a potential treatment for amblyopia: a mini-review. Vision Res. 2009 Oct;49(21):2535-49. doi: 10.1016/j.visres.2009.02.010. Epub 2009 Feb 27. PMID 19250947
- [Background] Mansouri B, Thompson B, Hess RF. Measurement of suprathreshold binocular interactions in amblyopia. Vision Res. 2008 Dec;48(28):2775-84. doi: 10.1016/j.visres.2008.09.002. Epub 2008 Nov 1. PMID 18809424
- [Background] Oscar A, Cherninkova S, Haykin V, Aroyo A, Levi A, Marinov N, Kostova S, Elenkov C, Veleva N, Chernodrinska V, Petkova I, Spitzer J. Amblyopia screening in Bulgaria. J Pediatr Ophthalmol Strabismus. 2014 Sep-Oct;51(5):284-8. doi: 10.3928/01913913-20140618-01. Epub 2014 Jun 25. PMID 24971584
- [Background] Scheiman MM, Hertle RW, Beck RW, Edwards AR, Birch E, Cotter SA, Crouch ER Jr, Cruz OA, Davitt BV, Donahue S, Holmes JM, Lyon DW, Repka MX, Sala NA, Silbert DI, Suh DW, Tamkins SM; Pediatric Eye Disease Investigator Group. Randomized trial of treatment of amblyopia in children aged 7 to 17 years. Arch Ophthalmol. 2005 Apr;123(4):437-47. doi: 10.1001/archopht.123.4.437. PMID 15824215
- [Background] Pizzorusso T, Medini P, Berardi N, Chierzi S, Fawcett JW, Maffei L. Reactivation of ocular dominance plasticity in the adult visual cortex. Science. 2002 Nov 8;298(5596):1248-51. doi: 10.1126/science.1072699. PMID 12424383
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- [Background] Stewart CE, Fielder AR, Stephens DA, Moseley MJ. Treatment of unilateral amblyopia: factors influencing visual outcome. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3152-60. doi: 10.1167/iovs.05-0357. PMID 16123414
- [Background] VON NOORDEN G. Principles of surgical treatment. Binocular vision and ocular motility. 1985:440-79.
- [Background] Abdelrazik ST, Khalil MF. Prevalence of amblyopia among children attending primary schools during the amblyogenic period in Minia county. Journal of the Egyptian Ophthalmological Society. 2014 Oct 1;107(4):220.
- [Background] Baker DH, Meese TS, Hess RF. Contrast masking in strabismic amblyopia: attenuation, noise, interocular suppression and binocular summation. Vision Res. 2008 Jul;48(15):1625-40. doi: 10.1016/j.visres.2008.04.017. Epub 2008 Jun 10. PMID 18547600
- [Background] Bi H, Zhang B, Tao X, Harwerth RS, Smith EL 3rd, Chino YM. Neuronal responses in visual area V2 (V2) of macaque monkeys with strabismic amblyopia. Cereb Cortex. 2011 Sep;21(9):2033-45. doi: 10.1093/cercor/bhq272. Epub 2011 Jan 24. PMID 21263036
- [Background] Foss AJ, Gregson RM, MacKeith D, Herbison N, Ash IM, Cobb SV, Eastgate RM, Hepburn T, Vivian A, Moore D, Haworth SM; I-BiT Steering group. Evaluation and development of a novel binocular treatment (I-BiT) system using video clips and interactive games to improve vision in children with amblyopia ('lazy eye'): study protocol for a randomised controlled trial. Trials. 2013 May 20;14:145. doi: 10.1186/1745-6215-14-145. PMID 23688108
- [Background] Hess RF, Mansouri B, Thompson B. A new binocular approach to the treatment of amblyopia in adults well beyond the critical period of visual development. Restor Neurol Neurosci. 2010;28(6):793-802. doi: 10.3233/RNN-2010-0550. PMID 21209494
- [Background] Hess RF, Thompson B, Baker DH. Binocular vision in amblyopia: structure, suppression and plasticity. Ophthalmic Physiol Opt. 2014 Mar;34(2):146-62. doi: 10.1111/opo.12123. PMID 24588532
- [Background] Maehara G, Thompson B, Mansouri B, Farivar R, Hess RF. The perceptual consequences of interocular suppression in amblyopia. Invest Ophthalmol Vis Sci. 2011 Nov 21;52(12):9011-7. doi: 10.1167/iovs.11-7748. PMID 22025565
- [Background] American Academy of Ophthalmology Basic and Clinical Science Course Subcommittee. Basic and Clinical Science Course. Pediatric Ophthalmology and Strabismus: Section 6. San Francisco, CA: American Academy of Ophthalmology. 2012.pp.61.
- [Background] Ophthalmology P. Strabismus Preferred Practice Pattern Panel. Amblyopia Preferred Practice Pattern Guidelines. San Francisco, CA: American Academy of Ophthamology. 2012
- [Background] Tsirlin I, Colpa L, Goltz HC, Wong AM. Behavioral Training as New Treatment for Adult Amblyopia: A Meta-Analysis and Systematic Review. Invest Ophthalmol Vis Sci. 2015 Jun;56(6):4061-75. doi: 10.1167/iovs.15-16583. PMID 26114483

DOCUMENTS (3):
  • Study Protocol (2022-11-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03255707/Prot_003.pdf
  • Statistical Analysis Plan (2022-11-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03255707/SAP_004.pdf
  • Informed Consent Form (2022-11-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT03255707/ICF_005.pdf